CLINICAL TRIAL: NCT06942949
Title: Evaluation of Enhanced Lithotripsy System (ELS) in the Treatment of Urinary Stones, A Pivotal Trial
Acronym: ELS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avvio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0002
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: Kidney Calculi; Ureteral Calculi
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- The ELS Trial is a prospective, multi-center, single arm study. (Experimental): All Subjects who qualify to participate in the ELS Trial will receive the experimental ELS procedure.
  Interventions: Device: ELS (Enhanced Lithotripsy System)

INTERVENTIONS:
Device: ELS (Enhanced Lithotripsy System) — ELS (Enhanced Lithotripsy System) utilizes low pressure ultrasound to actuate proprietary microbubbles administered into the urine to pit and fragment urinary stones.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the ELS to treat urinary stones. The ELS is intended to break urinary stones into small fragments that can pass during or after the procedure with less or no discomfort. Eligible patients are male or females, age 21 or older, with a single urinary stone in the ureter. Participants will undergo the ELS procedure and then be evaluated 30 days later for the presence or absence of urinary stone fragments on a CT scan. Subjects who still have stone present at Day 30 will be evaluated again at Day 60. Other outcome measures will be changes in pain, quality of life, and return to normal daily activities/work.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged >=21 Years
* Provides written informed consent
* One urinary stone within the ureter, size >=5 mm and <=10 mm present on CT
* Stone is indicated for Shock Wavve Lithotrips Per AUA 2026 guidelines
* Stone to be treated has a maximum density of <= 1200 HU

Exclusion Criteria:

* Anatomic presentations that would preclude obtaining an acoustic window for the ultrasound treatment
* Non-calcium based stones (e.g., uric acid stones)
* Untreated UTI
* Presence of abnormal skin conditions in the area to be treated
* Coagulation abnormality
* Inability to lay still for 30 minutes
* Pregnant
* Abnormal Kidney Function
* Any genitourinary history or procedure that has altered anatomy (e.g. urinary tract reconstruction)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | From ELS treatment to 30 Days afterward.
  CT assessment of the target stone demonstrating either (i) stone free status (zero fragments) or (ii) the presence of only stone fragments small enough to pass spontaneously (<=4 mm) at 30 Days post procedure.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Arizona State Urological Research Institute, Phoenix, Arizona
  - Michael G. Oefelein Clinical Trials, Bakersfield, California
  - San Diego Clinical Trials, La Mesa, California
  - Golden State Urology, Sacramento, California
  - University of Miami Hospital, Miami, Florida
  - Georgia Urology, Roswell, Georgia
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Wichita Urology Group, Wichita, Kansas
  - Minnesota Urology, Woodbury, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - SUNY - Upstate Medical University, Syracuse, New York
  - Duke, Durham, North Carolina
  - Urology San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Virginia Community Health, Culpeper, Virginia
  - Urology of Virginia, Virginia Beach, Virginia